CLINICAL TRIAL: NCT00200863
Title: Mechanism Underlying the Effects of Blue Light in Humans
Brief Title: Effects of Different Colors of Light on Human Physiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Steven W. Lockley, Neuroscientist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AT002129-01 (NIH); R01AT002129-01 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Healthy; Circadian Rhythm
Keywords: light; wavelength; action spectrum; circadian; melatonin; alertness; performance; arousal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): 420 nm light
  Interventions: Device: Monochromatic visible light exposure
- 2 (Experimental): 480 nm
  Interventions: Device: Monochromatic visible light exposure
- 3 (Experimental): 507 nm
  Interventions: Device: Monochromatic visible light exposure
- 4 (Experimental): 555 nm
  Interventions: Device: Monochromatic visible light exposure
- 5 (Experimental): 620 nm
  Interventions: Device: Monochromatic visible light exposure
- 6 (Experimental): 460 nm
  Interventions: Device: Monochromatic visible light exposure

INTERVENTIONS:
Device: Monochromatic visible light exposure — Monochromatic light in the visible range from 420-620 nm up to 60uW/cm2 for 6.5 hours

SUMMARY:
This study will determine which color of light is most effective in stimulating a range of biological functions in humans including activation of sleep-wake regulatory system (alertness, performance, microsleeps, brain activity), activation of the nervous system (heart rate, temperature, blood pressure, breathing rate), and shifting the timing of the internal 24-hour (circadian) pacemaker.

DETAILED DESCRIPTION:
Light has long been proposed to have a stimulatory effect on a range of biological functions in humans including increased feelings of activation, such as improved alertness or ability to perform. The mechanisms underlying how light stimulates these neurobiological systems remain to be elucidated. We propose to investigate the effects of different colors of light on human physiology, and in particular, test the claims that specific colors of light preferentially stimulate neurobiological, physiological and hormonal systems. Using classical photobiological techniques, we will construct action spectra for the effects of different colors of light on a range of non-image forming responses in humans.

We will test the hypotheses that: 1) light-induced activation of the neurobiological sleep-wake regulatory system, as indicated by increased alertness, faster reaction time, suppression of EEG alpha activity, microsleeps and slow rolling eye movements, and suppression of pineal melatonin, is most sensitive to retinal exposure to short wavelength blue light (460 nm) compared to equal photons of other colors of visible light; 2) light-induced activation of autonomic and hypothalamic-pituitary-adrenal axis measures of arousal, as indicated by increased heart rate variability, core body temperature, blood pressure, respiration rate, plasma cortisol levels and urinary catecholamines, is most sensitive to exposure to short wavelength blue light (460 nm) compared to equal photons of other colors; 3) phase shifts of the human circadian pacemaker, as assessed by changes in temperature, melatonin and cortisol rhythms, are most sensitive to exposure to short wavelength blue light (460 nm) compared to equal photons of other colors. The resultant action spectra will help to identify the photoreceptor mechanism(s) by which light activates arousal and circadian resetting, these non-image-forming physiological responses and enable us to distinguish between major candidate photoreceptive mechanisms, including potential novel photoreceptor systems, that might mediate such responses.

ELIGIBILITY:
Inclusion Criteria:

* Free from any acute, chronic or debilitating medical, psychological, or ophthalmological conditions
* Drug-free (including caffeine, nicotine, and alcohol) for entire study duration

Exclusion Criteria:

* History of drug or alcohol dependency
* History of psychiatric illnesses or evidence of psychopathology according to standardized questionnaires, or in a structured clinical interview
* Night shift work during the past 3 years
* Transmeridian travel in the last 3 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2005-04; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Subjective alertness prior to, during and after light exposure | 9.5 hours
Auditory psychomotor performance prior to, during and after light exposure | 9.5 hours
EEG power frequency prior to, during and after light exposure | 9.5 hours
Plasma melatonin and cortisol prior to, during and after light exposure | 60 hours
Heart rate, blood pressure, respiration rate and temperature prior to, during and after light exposure | 9.5 hours
Urinary catecholamines prior to, during and after light exposure | 32 hours

CONTACTS AND LOCATIONS:
Overall Officials: Steven W Lockley, Ph.D., Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Division of Sleep Medicine, Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Gooley JJ, Chamberlain K, Smith KA, Khalsa SB, Rajaratnam SM, Van Reen E, Zeitzer JM, Czeisler CA, Lockley SW. Exposure to room light before bedtime suppresses melatonin onset and shortens melatonin duration in humans. J Clin Endocrinol Metab. 2011 Mar;96(3):E463-72. doi: 10.1210/jc.2010-2098. Epub 2010 Dec 30. PMID 21193540